CLINICAL TRIAL: NCT01357759
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose-Escalation Trial of MORAb-022 in Healthy Subjects and Subjects With Rheumatoid Arthritis
Brief Title: Safety and Tolerability of MORAb-022 in Healthy and Rheumatoid Arthritis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MORAB022-001
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — gimsilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escalating doses of MORAb-022 (Experimental): Subjects with RA will be randomized into Cohorts 8 to 11, with each cohort consisting of five RA subjects per cohort (four active and one placebo).
  Interventions: Drug: MORAb-022
- Placebo (Placebo Comparator): Subjects with RA will be also randomized into Cohorts 8 to 11, with each cohort consisting of five RA subjects per cohort (four active and one placebo).
  Interventions: Drug: MORAb-022

INTERVENTIONS:
Drug: MORAb-022 — IV infusion of MORAb-022 at increasing doses starting with the minimal anticipated biological effect level (MABEL) which is 0.0085mg/kg.; IV infusion of Placebo (saline)
  Arms: Escalating doses of MORAb-022
Drug: MORAb-022 — IV infusion of MORAb-022 at increasing doses starting with the minimal anticipated biological effect level (MABEL) which is 0.0085mg/kg.; IV infusion of Placebo (saline)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-dose, dose escalation study in healthy male and or female subjects and subjects with Rheumatoid Arthritis (RA) to determine the safety and tolerability of MORAb-022.

ELIGIBILITY:
Inclusion Criteria for Rheumatoid Arthritis (RA) Subjects:

* Male or female subjects age greater than or equal to 18 years and less than or equal to 75 years.
* Subjects with RA diagnosis per the 2010 Rheumatoid Arthritis Classification Criteria per American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR.)
* BMI less than or equal to 35 kg/m2 at Screening.
* Active RA characterized by DAS28 score of less than or equal to 5.1 at Screening.
* Have been stabilized on their current dose (up to 25 mg/week) of methotrexate(MTX) for at least 4 weeks before randomization.

Exclusion Criteria for Rheumatoid Arthritis (RA)Subjects:

* Subjects with severe active RA and are not on a stable therapeutic regimen at Screening.
* Subjects without significant articular RA.
* Relevant history of significant respiratory disease (e.g., chronic bronchitis, asthma in last 5 years, chronic obstructive pulmonary disease, tuberculosis, interstitial lung disease, such as pneumonitis and pulmonary alveolar proteinosis, as well as significant inhalation exposure to silicon and other substances) that required treatment and/or follow up under the direction of a physician.
* Presence of GM-CSF autoantibodies above normal at Screening.
* Abnormal chest x-ray or PFTs as judged by the investigator at Screening as clinically significant.
* Positive Quantiferon test.
* History of clinically relevant hypersensitivity reactions (e.g., to gold therapy)
* History of medication use that might have carryover effects during the study.
* Previous administration of a GM-CSF modulator within 6 months of randomization, or previous administration of a monoclonal antibody or immunoglobulin fusion protein that is not (or worded as "other than") a GM-CSF modulator within 3 months of randomization.
* Use of any biological therapy other than the test article during the study (informed consent to termination visit)
* Subjects who consume greater than 14 alcoholic drinks per week for males or 7 alcoholic drinks per week for females.
* Weight greater than 120 kg at Screening.
* Use of parenteral and/or intra-articular steroids, immunosuppressants, investigational drugs, and oral anticoagulant drugs within 4 weeks prior to randomization. Oral steroid treatment is permitted if the dosage is less than or equal to 10 mg of prednisone daily, is stable for a minimum of 4 weeks before the study and remains unchanged throughout the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety to measures to include adverse events, clinical laboratory results, vital signs, ECGs, physical examinations, local tolerability at the infusion site single escalating intravenous (IV) doses of MORAb-022 in healthy subjects and subjects with RA. | Approximately 113 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan J. Kivitz, MD, CPI, Principal Investigator — Altoona Center for Clinical Research; Lydie Hazan, MD, Principal Investigator — Axis Clinical Trials; Chrysoula Pappa, MD, Principal Investigator — Seaview Jacksonville, LLC; William M Schnitz, MD, Principal Investigator — Lynn Health Science Institute
Locations (5):
- United States (4):
  - Axis Clinical Trials, Los Angeles, California
  - Seaview Jacksonville, LLC, Jacksonville, Florida
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
- Pharmaceutical Research Associates Group B.V., Zuidlaren, Netherlands